CLINICAL TRIAL: NCT02912208
Title: Eltrombopag for the Treatment of Thrombocytopenia Due to Low- and Intermediate Risk Myelodysplastic Syndromes (EQoL-MDS)
Brief Title: Eltrombopag for the Treatment of Thrombocytopenia Due to Low- and Intermediate Risk Myelodysplastic Syndromes
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Associazione Qol-one (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EQoL-MDS
Record Dates: First submitted 2016-09-09; First posted 2016-09-23 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Myelodysplastic Syndromes; Thrombocytopenia
MeSH Terms: conditions — Myelodysplastic Syndromes; Thrombocytopenia | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Eltrombopag) (Experimental): Arm 1 is the active treatment arm
  Interventions: Drug: Eltrombopag/Revolade
- Arm 2 (Placebo) (Placebo Comparator): Arm 2 is the control arm
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Eltrombopag/Revolade — Eltrombopag 50 mg once daily has been selected as the starting dose for this study. Thereafter, dependent on platelet response the dose of study medication can be increased by 50 mg every 2 weeks, up to a maximum dose of 300 mg once daily (150 mg in subjects of East Asian ethnicity).
  Arms: Arm 1 (Eltrombopag)
Other: Placebo — The administration is the same of eltrombopag
  Arms: Arm 2 (Placebo)

SUMMARY:
Myelodysplastic syndromes (MDS) prevail in older age and are characterized by ineffective erythropoiesis and peripheral cytopenias. Supportive therapy is the main therapeutic option for most patients. Quality of Life (QoL) is mainly deteriorated by anemia and by the limitations associated with thrombocytopenia, neutropenia and transfusion dependence. The only available treatment for severe thrombocytopenia, in the presence of bleeding, is platelet transfusion.

Eltrombopag is an orally bioavailable agonist of the thrombopoietin receptor. In adult patients with chronic immune thrombocytopenia (ITP), Eltrombopag rapidly increases platelet counts and significantly reduces bleeding episodes during treatment. Eltrombopag is well tolerated. In 2007, Eltrombopag has received the Orphan Drug Designation for the treatment of ITP (EMEA/OD/031/07), and in 2008 the Food and Drug Association approved Eltrombopag for the treatment of ITP refractory or resistant. It has been shown that in patients affected by MDS and by acute myeloid leukemia, Eltrombopag neither increases the proliferation, nor the clonogenic growth capacity of bone marrow blasts. Furthermore, Eltrombopag induces an increase in the megakaryocytic differentiation and in the formation of normal megakaryocytic colonies. These results provide the rationale for pursuing further research on Eltrombopag for the treatment of thrombocytopenia in case of MDS.

The study is open to adult patients with myelodysplastic syndrome (MDS) with thrombocytopenia and low- or intermediate-1 IPSS risk (Index Prognostic Score System).

Severe thrombocytopenia associated with MDS may lead to death from hemorrhage, even in low prognostic risk patients. The benefit of platelet transfusion is short-termed. Patients become refractory in the long term. The availability of a treatment that induces the increase of platelet count is extremely important, either in terms of quality of life, and in overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (18 years of age or older) with low or intermediate-1 IPSS risk MDS and stable disease.
2. Subjects must have a platelet count taken within the 4 weeks prior to randomization that is <30 Gi/L.
3. Subjects must be ineligible or relapsed or refractory to receive other treatment options (such as azacitidine or lenalidomide) and must be ineligible to receive intensive chemotherapy or autologous/allogeneic stem cell transplantation.
4. Subjects must have platelet count and platelet transfusion data available over a period of 8 weeks prior to randomization.
5. During the 2 months prior to randomization, subjects must have a baseline Bone Marrow examination which includes cytomorphology and cytogenetics. Histopathology should be performed.
6. Erythropoiesis-stimulating agents (ESAs) in anemic subjects or granulocyte colonystimulating factor (G-CSF) in subjects with severe neutropenia and recurrent infections are allowed during the study as per accepted standards. Subjects who enter the study on ESAs or G-CSF should continue at the same dose schedule until the optimal dose of study medication has been established.
7. ECOG (Eastern Cooperative Oncology Group) Performance Status 0-3
8. Subject is able to understand and comply with protocol requirements and instructions.
9. Subject has signed and dated informed consent.
10. Adequate baseline organ function defined by the criteria below:

    total bilirubin (except for Gilbert's Syndrome) ≤ 1.5 x Upper Limit Normal Alanine aminotransferase and Aspartate aminotransferase ≤ 3 x Upper Limit Normal creatinine ≤ 2 x Upper Limit Normal albumin must not be below the lower limit of normal by more than 20%.
11. Subject is practicing an acceptable method of contraception. Female subjects (or female partners of male subjects) must either be of non-childbearing potential (hysterectomy, bilateral oophorectomy, bilateral tubal ligation or post-menopausal >1 year), or of childbearing potential and use of an highly effective method of contraception from 2 weeks prior to administration of study medication, throughout the study, and 28 days after completion or premature discontinuation from the study.

Exclusion Criteria:

1. MDS with intermediate-2 or high IPSS risk.
2. History of treatment for cancer other than MDS with systemic chemotherapy and/or radiotherapy within the last 2 years.
3. History of treatment with romiplostim or other Thrombopoietin receptor agonists.
4. Pre-existing cardiovascular disease (including congestive heart failure, New York Heart Association Grade III/IV), or arrhythmia known to increase the risk of thromboembolic events (e.g. persistent atrial fibrillation), or subjects with a QTc >450 msec (QTc >480 msec for subjects with Bundle Branch Block).
5. BM fibrosis that leads to an inability to aspirate marrow for assessment.
6. Peripheral monocytosis > 1000/uL prior to Day 1 of study medication.
7. Leukocytosis >=25,000/uL prior to Day 1 of study medication.
8. Female subjects who are nursing or pregnant (positive serum or urine Beta-human chorionic gonadotropin [B-hCG] pregnancy test) at screening or pre-dose on Day 1.
9. Current alcohol or drug abuse.
10. Treatment with an Investigational Product within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
11. Active and uncontrolled infections.
12. Subjects infected with Hepatitis B, C or Human Immunodeficiency Virus (HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2011-06-11 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Response rate | Six months
  Proportion of patients achieving a complete response (CR) or response (R) during the treatment period
Safety and Tolerability (number of adverse events) | Six month
  Safety and tolerability in terms of frequency of adverse events (AE) and serious adverse events (SAE)
Duration of platelet response | five years
long-term safety and tolerability (number adverse events in the long term) | five years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 and number of adverse events reporting in accordance with CTCAE v4.0

SECONDARY OUTCOMES:
Quality of life (QoL) score | six months
  to evaluate the changes of the quality of life in the two arms
number of monthly platelet transfusions | six months
duration of transfusion independence | six months
time to response | six months
  time to response (time from starting treatment to time of achievement of CR or PR)
incidence and severity of bleeding | six months
  incidence and severity of bleeding using the WHO (World Health Organization)Bleeding Scale
overall survival | 2 and 5 years
  overall survival (OS) at 2 and at 5 years
leukemia-free survival (LFS) | 2 and 5 years
  leukemia-free survival (LFS) at 2 and at 5 years (events for LFS are defined as death and progression to AML);

CONTACTS AND LOCATIONS:
Overall Officials: Esther Natalie Oliva, Study Chair — QOL-ONE Associazione Culturale e di Ricerca
Locations (64):
- France (22):
  - CHU Amiens, Amiens
  - Centre d'Avignon, Avignon
  - Hôpital de la Côte Basque, Bayonne
  - Centre d'Avicenne, Hôpital d'Avicenne, Bobigny
  - CHU de Haut-Lévèque, Bordeaux
  - Centre Hospitalier de Boulogne Sur Mer, Boulogne-sur-Mer
  - CHU Clémenceau, Caen
  - Centre Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - Centre Le Mans, Le Mans
  - Hôpital Saint Vincent de Paul, Lille
  - CHRU de Limoges, Limoges
  - Centre de Marseille, Marseille
  - CHU Brabois, Nancy
  - Centre de Nantes, Nantes
  - Hopital Archet 1, Nice
  - Centre Hospitalier Universitaire de Nimes, Nîmes
  - Centre de St Louis, Hôpital St Louis, Paris
  - Centre Hospitalier de la Région d'Annecy, Pringy
  - Centre de Rouen, Centre Henri Becquerel, Rouen
  - CHU Purpan, Toulouse
  - CHU de Bretonneau, Tours
- Germany (2):
  - Heinrich-Heine-Universität Düsseldorf, Düsseldorf
  - Universitätsmedizin Mannheim, Mannheim
- Italy (33):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo, Alessandria, AL
  - Ospedale Riuniti, Ancona, AN
  - Ospedale Cardinal Massaia, Asti, AT
  - A.O. S. Giovanni Moscati, Avellino, AV
  - Policlinico Università di Bari, Bari, BA
  - Ospedale A. Perrino, Brindisi, BR
  - Ospedale "Roberto Binaghi", Cagliari, CA
  - Ospedale L'Annunziata, Cosenza, CS
  - Ospedale Ferrarotto, Catania, CT
  - Ospedale Garibaldi, Catania, CT
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, FG
  - Azienda Ospedaliera Universitaria Careggi, Florence, FI
  - Università degli Studi di Genova, Genova, GE
  - Ospedale Vito Fazzi, Lecce, LE
  - IRCCS Ospedale Maggiore Policlinico, Milan, MI
  - Ospedale Niguarda, Milan, MI
  - Ospedale Civile Spirito Santo, Pescara, PE
  - Azienda Ospedaliera Bianchi-Melacrino-Morelli, Reggio Calabria, RC
  - Arcispedale di Santa Maria Nuova, Reggio Emilia, RE
  - A.O. San Camillo Forlanini, Roma, RM
  - Ospedale Sant'Eugenio, Roma, RM
  - Policlinico Agostino Gemelli, Roma, RM
  - Università Campus Bio Medico di Roma, Roma, RM
  - Azienda Ospedaliera Sant'Andrea, Rome, RM
  - IRCCS Istituto Regina Elena, Rome, RM
  - Ospedale Nuova Regina Margherita, Rome, RM
  - Policlinico Umberto I, Rome, RM
  - Policlinico Universitario Tor Vergata, Rome, RM
  - A.O.U. San Giovanni di Dio e Ruggì D'Aragona, Salerno, SA
  - Policlinico Santa Maria alle Scotte, Siena, SI
  - A.O. Santa Maria, Terni, TE
  - A.O. Citta' della Salute e della Scienza di Torino, Torino, TO
  - U.O. Citta' della Salute e della Scienza di Torino, Torino, TO
- Slovenia (7):
  - General Hospital Celje, Celje
  - Univerzitetni klinini center Ljubljana, Ljubljana
  - University Medical Centre Maribor, Maribor
  - General Hospital Murska Sobota, Murska Sobota
  - General Hospital Nova Gorica, Nova Gorica
  - General Hospital Novo mesto, Novo Mesto
  - General Hospital Slovenj Gradec, Slovenj Gradec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oliva EN, Riva M, Niscola P, Santini V, Breccia M, Giai V, Poloni A, Patriarca A, Crisa E, Capodanno I, Salutari P, Reda G, Cascavilla N, Ferrero D, Guarini A, Tripepi G, Ianni G, Russo E, Castelli A, Fattizzo B, Beltrami G, Bocchia M, Molteni A, Fenaux P, Germing U, Ricco A, Palumbo GA, Impera S, Di Renzo N, Rivellini F, Buccisano F, Stamatoullas-Bastard A, Liberati AM, Candoni A, Delfino IM, Arcadi MT, Cufari P, Rizzo L, Bova I, D'Errigo MG, Zini G, Latagliata R. Eltrombopag for Low-Risk Myelodysplastic Syndromes With Thrombocytopenia: Interim Results of a Phase II, Randomized, Placebo-Controlled Clinical Trial (EQOL-MDS). J Clin Oncol. 2023 Oct 1;41(28):4486-4496. doi: 10.1200/JCO.22.02699. Epub 2023 Jun 9. PMID 37294914